CLINICAL TRIAL: NCT02403115
Title: Validation of the Assay of Circulating Antibodies Against Glomerular Neo-autoantigens as a Surrogate Biomarker of the Development of Lupus Nephritis
Brief Title: Prediction of Outcome of Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, MD, Istituto Giannina Gaslini
Other Study IDs: SLE1
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Lupus Nephritis: Collection of serum at onset and during subsequent follow-up at 6, 12, 24 and 36 months for the dosage of circulating autoantibodies.
  Interventions: Other: Serum collection
- Incident SLE without nephritis: Collection of serum at onset and during subsequent follow-up at 6, 12, 24 and 36 months for the dosage of circulating autoantibodies, in order to evaluate the presence of nephritic manifestations.
  Interventions: Other: Serum collection
- Prevalent SLE without nephritis: Collection of serum at onset and during subsequent follow-up at 6, 12, 24 and 36 months for the dosage of circulating autoantibodies in order to evaluate the presence of nephritic manifestations.
  Interventions: Other: Serum collection
- Rheumatoid arthritis: Collection of serum at onset and during subsequent follow-up at 6, 12, 24 and 36 months for the dosage of circulating autoantibodies in order to evaluate the presence of nephritic manifestations.
  Interventions: Other: Serum collection
- Membranous glomerulonephritis: Collection of serum at onset and during subsequent follow-up at 6, 12, 24 and 36 months for the dosage of circulating autoantibodies in order to exclude secondary forms of the disease.
  Interventions: Other: Serum collection

INTERVENTIONS:
Other: Serum collection — Clinical tests (renal function, complete blood count, CRP, ANA, dsDNA, urinalysis) will be performed at fixed time intervals (6, 12, 24 and 36 months) and the surplus of blood sample will form the serum bank used for the study

SUMMARY:
The purpose of this study is to clarify the mechanisms involved in the formation and glomerular deposition of immune complexes in lupus nephritis.

The determination of an antibody pattern specific for systemic lupus erythematosus and lupus nephritis may also have a role in predicting disease progression in patients with systemic lupus erythematosus without renal impairment. As for the patients enrolled in the study, the determination of their antibody patterns may contribute to a more targeted and personalized treatment, allowing a prediction of disease progression and the introduction of early targeted treatments, in order to block the onset and/or progression of renal damage.

DETAILED DESCRIPTION:
Prospective multicenter study on the validity of levels of circulating antibodies to glomerular neo-autoantigens (alpha-enolase and annexin AI) and implantable antigens (anti-DNA, histone, istone3, istone4, C1q) as a surrogate biomarker for the diagnosis of lupus nephritis.

The study will involve the collection of serum from patients with lupus nephritis at onset and during subsequent follow-up at 6, 12, 24 and 36 months for the titration of circulating autoantibodies.

As a control the investigators will use the sera of patients with systemic lupus erythematosus without nephropathy, collected at the same time intervals.

The investigators will also assess the antibody positivity in groups of patients with rheumatologic disease similar to lupus (rheumatoid arthritis) and in patients with autoimmune nephropathy without extrarenal clinical signs.

Regarding patients with systemic lupus erythematosus the investigators will collect sera of both incident and prevalent patients in order to monitor changes in antibody levels in conjunction with the development of renal disease.

Clinical tests (renal function, complete blood count, C reactive protein (CRP), ANA, native DNA (nDNA), urine analysis) will be performed at 6, 12, 24 and 36 months and the surplus of blood samples will be used to create the serum bank of the study.

Samples will be collected in the pediatric nephrology of Giannina Gaslini Children Hospital, Genoa (coordinator centre) and in 5 rheumatological (Genoa, Pisa, Pavia, Padova, Brescia) and 6 nephrological (Milan, Genoa, Parma, Brescia, Bologna and Reggio Emilia) italian adults departments .

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 65 years
* Diagnosis of lupus nephritis-systemic lupus erythematosus (systemic lupus erythematosus, rheumatoid arthritis and membranous nephropathy for controls)
* Informed consent

Exclusion Criteria:

* Severe infections in place
* Malignancies of any current or history
* Chronic hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) positive
* Breast-feeding or pregnant
* Known hypersensitivity to drugs

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * 250 patients with newly diagnosed lupus nephritis (stage I-VI according to WHO classification). First serum will be collected at the time of renal biopsy (study group).
  * 250 patients with incident or prevalent systemic lupus erythematosus (according to ARA criteria) and no signs of nephropathy (control group).
  * 50 patients with rheumatoid arthritis (according to ARA criteria), without documented nephropathy (control group)
  * 250 patients with histological diagnosis of membranous nephropathy (control group).
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Proteinuria at 12, 24 and 36 months | 12, 24, 36 months
  proteinuria measured on a 24-hour urine collection.

SECONDARY OUTCOMES:
Renal function | 36 months
  estimated glomerular filtration rate (eGFR) measured according to Revised Bedside Schwartz Formula (4-17 years old patients) or CKD-EPI Creatinine 2009 Equation (18-64 years old patients)

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco Ghiggeri, MD, Study Director — IRCCS Giannina Gaslini, Genoa
Locations (1):
- IRCCS Giannina Gaslini Children Hospital, Genoa, Italy/GE, Italy

REFERENCES:
- [Background] Cameron JS. Lupus nephritis. J Am Soc Nephrol. 1999 Feb;10(2):413-24. doi: 10.1681/ASN.V102413. No abstract available. PMID 10215343
- [Background] Yu C, Gershwin ME, Chang C. Diagnostic criteria for systemic lupus erythematosus: a critical review. J Autoimmun. 2014 Feb-Mar;48-49:10-3. doi: 10.1016/j.jaut.2014.01.004. Epub 2014 Jan 21. PMID 24461385
- [Background] Madaio MP. The relevance of antigen binding to the pathogenicity of lupus autoantibodies. Kidney Int. 2012 Jul;82(2):125-7. doi: 10.1038/ki.2012.159. PMID 22743561
- [Background] Waldman M, Madaio MP. Pathogenic autoantibodies in lupus nephritis. Lupus. 2005;14(1):19-24. doi: 10.1191/0961203305lu2054oa. PMID 15732283
- [Background] Bagavant H, Fu SM. Pathogenesis of kidney disease in systemic lupus erythematosus. Curr Opin Rheumatol. 2009 Sep;21(5):489-94. doi: 10.1097/BOR.0b013e32832efff1. PMID 19584729
- [Background] Hanrotel-Saliou C, Segalen I, Le Meur Y, Youinou P, Renaudineau Y. Glomerular antibodies in lupus nephritis. Clin Rev Allergy Immunol. 2011 Jun;40(3):151-8. doi: 10.1007/s12016-010-8204-4. PMID 20414746
- [Background] Kramers C, Hylkema MN, van Bruggen MC, van de Lagemaat R, Dijkman HB, Assmann KJ, Smeenk RJ, Berden JH. Anti-nucleosome antibodies complexed to nucleosomal antigens show anti-DNA reactivity and bind to rat glomerular basement membrane in vivo. J Clin Invest. 1994 Aug;94(2):568-77. doi: 10.1172/JCI117371. PMID 8040312
- [Result] Bruschi M, Galetti M, Sinico RA, Moroni G, Bonanni A, Radice A, Tincani A, Pratesi F, Migliorini P, Murtas C, Franceschini F, Trezzi B, Brunini F, Gatti R, Tardanico R, Barbano G, Piaggio G, Messa P, Ravani P, Scolari F, Candiano G, Martini A, Allegri L, Ghiggeri GM. Glomerular Autoimmune Multicomponents of Human Lupus Nephritis In Vivo (2): Planted Antigens. J Am Soc Nephrol. 2015 Aug;26(8):1905-24. doi: 10.1681/ASN.2014050493. Epub 2014 Nov 14. PMID 25398787
- [Result] Bruschi M, Sinico RA, Moroni G, Pratesi F, Migliorini P, Galetti M, Murtas C, Tincani A, Madaio M, Radice A, Franceschini F, Trezzi B, Bianchi L, Giallongo A, Gatti R, Tardanico R, Scaloni A, D'Ambrosio C, Carnevali ML, Messa P, Ravani P, Barbano G, Bianco B, Bonanni A, Scolari F, Martini A, Candiano G, Allegri L, Ghiggeri GM. Glomerular autoimmune multicomponents of human lupus nephritis in vivo: alpha-enolase and annexin AI. J Am Soc Nephrol. 2014 Nov;25(11):2483-98. doi: 10.1681/ASN.2013090987. Epub 2014 May 1. PMID 24790181
- [Derived] Angeletti A, Bruschi M, Moroni G, Sinico RA, Franceschini F, Fredi M, Vaglio A, Cavagna L, Petretto A, Pratesi F, Migliorini P, Locatelli F, Pazzola G, Pesce G, Bagnasco M, Manfredi A, Ramirez GA, Esposito P, Murdaca G, Negrini S, Cipriani L, Trezzi B, Emmi G, Cavazzana I, Binda V, d'Alessandro M, Fenaroli P, Pisani I, Garibotto G, Montecucco C, Santoro D, Scolari F, Volpi S, Mosca M, Tincani A, Candiano G, Prunotto M, Verrina E, Ravelli A, Ghiggeri GM. Second Wave Antibodies in Autoimmune Renal Diseases: The Case of Lupus Nephritis. J Am Soc Nephrol. 2021 Dec 1;32(12):3020-3023. doi: 10.1681/ASN.2021050659. Epub 2021 Dec 1. PMID 34599042
- [Derived] Bruschi M, Moroni G, Sinico RA, Franceschini F, Fredi M, Vaglio A, Cavagna L, Petretto A, Pratesi F, Migliorini P, Manfredi A, Ramirez GA, Esposito P, Negrini S, Trezzi B, Emmi G, Santoro D, Scolari F, Volpi S, Mosca M, Tincani A, Candiano G, Prunotto M, Verrina E, Angeletti A, Ravelli A, Ghiggeri GM. Neutrophil Extracellular Traps in the Autoimmunity Context. Front Med (Lausanne). 2021 Mar 22;8:614829. doi: 10.3389/fmed.2021.614829. eCollection 2021. PMID 33829021
- [Derived] Bruschi M, Moroni G, Sinico RA, Franceschini F, Fredi M, Vaglio A, Cavagna L, Petretto A, Pratesi F, Migliorini P, Locatelli F, Pazzola G, Pesce G, Bagnasco M, Manfredi A, Ramirez GA, Esposito P, Murdaca G, Negrini S, Cipriani L, Trezzi B, Emmi G, Cavazzana I, Binda V, Fenaroli P, Pisani I, Garibotto G, Montecucco C, Santoro D, Scolari F, Mosca M, Tincani A, Candiano G, Prunotto M, Volpi S, Verrina E, Angeletti A, Ravelli A, Ghiggeri GM. Serum IgG2 antibody multicomposition in systemic lupus erythematosus and lupus nephritis (Part 1): cross-sectional analysis. Rheumatology (Oxford). 2021 Jul 1;60(7):3176-3188. doi: 10.1093/rheumatology/keaa767. PMID 33374003
- [Derived] Bruschi M, Moroni G, Sinico RA, Franceschini F, Fredi M, Vaglio A, Cavagna L, Petretto A, Pratesi F, Migliorini P, Locatelli F, Pazzola G, Pesce G, Bagnasco M, Manfredi A, Ramirez GA, Esposito P, Murdaca G, Negrini S, Cipriani L, Trezzi B, Emmi G, Cavazzana I, Binda V, d'Alessandro M, Fenaroli P, Pisani I, Garibotto G, Montecucco C, Santoro D, Scolari F, Volpi S, Mosca M, Tincani A, Candiano G, Prunotto M, Verrina E, Angeletti A, Ravelli A, Ghiggeri GM. Serum IgG2 antibody multi-composition in systemic lupus erythematosus and in lupus nephritis (Part 2): prospective study. Rheumatology (Oxford). 2021 Jul 1;60(7):3388-3397. doi: 10.1093/rheumatology/keaa793. PMID 33351137
- [Derived] Bruschi M, Bonanni A, Petretto A, Vaglio A, Pratesi F, Santucci L, Migliorini P, Bertelli R, Galetti M, Belletti S, Cavagna L, Moroni G, Franceschini F, Fredi M, Pazzola G, Allegri L, Sinico RA, Pesce G, Bagnasco M, Manfredi A, Ramirez GA, Ramoino P, Bianchini P, Puppo F, Pupo F, Negrini S, Mattana F, Emmi G, Garibotto G, Santoro D, Scolari F, Ravelli A, Tincani A, Cravedi P, Volpi S, Candiano G, Ghiggeri GM. Neutrophil Extracellular Traps Profiles in Patients with Incident Systemic Lupus Erythematosus and Lupus Nephritis. J Rheumatol. 2020 Mar;47(3):377-386. doi: 10.3899/jrheum.181232. Epub 2019 May 15. PMID 31092713